CLINICAL TRIAL: NCT02723435
Title: An Open-Label Extension Study of Post-Transplant Maintenance Midostaurin (PKC412) in Elderly Patients (Age ≥ 60 Years) With FLT3-ITD/TKD Mutated AML Who Previously Received Midostaurin and Decitabine as Part of Study HEMAML0022 / CPKC412AUS27T
Brief Title: Midostaurin in Treating Older Patients With Mutated Acute Myeloid Leukemia Post-Transplant
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Logistical and administrative issues
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, David Iberri, Clinical Assistant Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-31582; NCI-2016-00424 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HEMAML0022-EXT (Other: OnCore); NCT02723435 (Other: Stanford University)
Record Dates: First submitted 2016-03-25; First posted 2016-03-30 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Acute Myeloid Leukemia With Gene Mutations; Adult Acute Myeloid Leukemia in Remission
MeSH Terms: interventions — midostaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Midostaurin (Experimental): Beginning 30 days post-HCT, participants receive oral midostaurin twice-a-day in 28-day treatment cycles, continuing up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Midostaurin

INTERVENTIONS:
Drug: Midostaurin — Given PO
  Other Names: Rydapt; CGP 41251; N-benzoyl-staurosporine; PKC-412

SUMMARY:
This phase 2 trial studies the side effects and how well midostaurin works in treating older patients with acute myeloid leukemia with change in genetic material post-hematopoietic cell transplantation. Midostaruin may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving midostaruin post-transplant may improve patient outcomes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy and safety of maintenance midostaurin (a fms related tyrosine kinase 3 [FLT3] inhibitor) for elderly patients with FLT3-internal tandem duplication (ITD)/tyrosine kinase domain (TKD) mutated acute myeloid leukemia (AML) who were previously enrolled on study HEMAML0022/CPKC412AUS27T and have then undergone allogeneic transplant.

SECONDARY OBJECTIVES:

I. To determine whether maintenance midostaurin after allogeneic transplant decreases the relapse rate in patients with FLT3-ITD/TKD mutated AML.

OUTLINE:

Beginning 30 days post-hematopoietic cell transplantation (HCT), patients receive midostaurin orally (PO) twice daily (BID) on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then up to 1 year.

ELIGIBILITY:
INCLUSION CRITERIA

* Elderly patients with FLT3-mutated acute myeloid leukemia (AML)
* Prior enrollment in Stanford study IRB-25737
* In continued complete remission
* ≥ 30 days but ≤ 90 days post allogeneic hematopoietic cell transplant (HCT); treatment on this study protocol must begin before day 90 post-HCT
* Absolute neutrophil count (ANC) ≥ 1000 cells/uL
* Hemoglobin ≥ 8.0 g/dL and not requiring regular transfusions
* Platelets ≥ 50,000 cells/uL and not requiring regular transfusions
* Aspartate aminotransferase (AST) ≤ 2.5 times upper limit of normal (ULN)
* Alanine aminotransferase (ALT) ≤ 2.5 X ULN
* Serum bilirubin ≤ 2.5 times ULN
* Ability to give written informed consent, including via legally authorized representative
* Corrected QT (QTc) ≤ 450 msec
* Ejection fraction (EF) ≥ 45% by 2-dimensional transthoracic echocardiography (TTE) or multiple-gated acquisition (MUGA)
* Sexually active males, including vasectomized males, must agree via informed consent to use a condom during vaginal, anal, or oral intercourse, while taking midostaurin and for 5 months after stopping midostaurin
* Females must have or be:

  * Negative pregnancy test, within 21 days of the first dose of midostaurin OR
  * Not of childbearing potential as follows:

    * Has undergone a hysterectomy or bilateral oophorectomy;
    * Has not had menses at any time in the preceding 24 consecutive months

EXCLUSION CRITERIA

* Uncontrolled acute graft-vs-host disease (GVHD) grade 3 to 4
* Uncontrolled active infection
* Evidence of active AML (eg, circulating peripheral blasts on complete blood count)
* Known confirmed diagnosis of human immunodeficiency virus (HIV) infection
* Known confirmed diagnosis of active viral hepatitis
* QTc > 450 msec
* Congenital long QT syndrome
* History of presence of sustained ventricular tachycardia, history of ventricular fibrillation or torsades de pointes
* Bradycardia defined as heart rate (HR) < 50 beats per minute (bpm)
* Bifascicular block (right bundle branch block plus left anterior hemiblock)
* Congestive heart failure (CHF) New York Heart Association (NYHA) class 3 or 4
* Cardiac ejection fraction (EF) < 45% within 28 days prior to starting cycle 1
* Other known malignancy (except carcinoma in situ)
* Other concurrent severe and/or uncontrolled medical condition which could compromise participation in the study, eg:

  * Uncontrolled diabetes
  * Chronic active pancreatitis
  * Myocardial infarction within 6 months
  * Poorly-controlled hypertension
  * Chronic kidney disease
* Received any investigational agent within 30 days prior to day 1
* Antineoplastic chemotherapy or radiotherapy within 28 days prior to cycle 1
* No plans for concurrent chemotherapy while on study (exception: antineoplastic drugs used as part of GVHD prophylaxis or treatment)
* Any surgical procedure, excluding central venous catheter placement, bone marrow biopsy or other minor procedures (eg, skin biopsy) within 14 days of day 1
* Unwillingness or inability to comply with the protocol
* Known malignant disease of the central nervous system
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to midostaurin
* Concomitant use of strong inhibitors of cytochrome P450 family 3 subfamily A member 4 (CYP3A4)
* Pregnant or lactating
* Women of child-bearing potential

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Event-free survival | Up to 1 year
Incidence of adverse events using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 30 days
Overall survival | Up to 1 year
  Calculated and reported with Kaplan Meier curves. The statistical analyses will focus on estimation rather than hypothesis testing. Two-sided 95% confidence intervals will be presented, using the Clopper-Pearson method for proportions and using Greenwood's formula for time to event outcomes.
Relapse free survival | Up to 1 year
  Calculated and reported with Kaplan Meier curves. The statistical analyses will focus on estimation rather than hypothesis testing. Two-sided 95% confidence intervals will be presented, using the Clopper-Pearson method for proportions and using Greenwood's formula for time to event outcomes.

SECONDARY OUTCOMES:
Relapse rate after allogeneic transplant | Up to 1 year
  Described using proportions.

CONTACTS AND LOCATIONS:
Overall Officials: David Iberri, MD, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No